CLINICAL TRIAL: NCT03614663
Title: A Randomized, Double-Blind, Placebo-Controlled Multiple-Center, Efficacy and Safety Study of ZYN002 Administered as a Transdermal Gel to Children and Adolescents With Fragile X Syndrome
Brief Title: Clinical Study Of caNNabidiol in childrEn and adolesCenTs With Fragile X (CONNECT-FX)
Acronym: CONNECT-FX
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zynerba Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZYN2-CL-016
Record Dates: First submitted 2018-07-10; First posted 2018-08-03 (Actual); Results first posted 2022-06-16 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2020-07

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ZYN002 - Cannabidiol transdermal gel (Experimental): ZYN002 supplied as a transdermal gel. Patients weighing less than or equal to 35 kg will be randomized to receive either 125 mg cannabidiol Q12H or placebo.
  Patients weighing greater than 35 kg will be randomized to receive 250 mg cannabidiol Q12H or placebo.
  Interventions: Drug: ZYN002 - Cannabidiol Transdermal Gel
- Placebo transdermal gel (Placebo Comparator): Matching ZYN002 placebo supplied as a transdermal gel.
  Interventions: Other: Placebo Transdermal Gel

INTERVENTIONS:
Drug: ZYN002 - Cannabidiol Transdermal Gel — Pharmaceutically manufactured. Cannabidiol formulated as a clear gel (transdermal delivery)
  Arms: ZYN002 - Cannabidiol transdermal gel
Other: Placebo Transdermal Gel — Placebo formulated as a clear gel (transdermal delivery)
  Other Names: Placebo Comparator; Matching Placebo
  Arms: Placebo transdermal gel

SUMMARY:
This trial will evaluate the efficacy and safety of ZYN002, a clear cannabidiol gel that can be applied to the skin (called transdermal application) twice a day for the treatment of behavioral symptoms of Fragile X Syndrome (FXS). Eligible participants will then participate in up to a 14 week treatment period, where all participants will receive placebo or active study drug. Patients ages 3 to < 18 years, will be eligible to participate.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multiple-center study, to assess the efficacy and safety of ZYN002, a pharmaceutically manufactured cannabidiol, formulated as a transdermal gel, for the treatment of children and adolescent with FXS. Approximately 204 male and female patients, ages 3 to < 18 years, will undergo a screening process. Eligible participants will be randomized 1:1 to either trial drug or placebo and will undergo a 14-week treatment period. Randomization will be stratified by gender, weight category and geographic region. All participants may receive placebo during the trial. Participants who are taking anti-seizure drugs may undergo an additional 1-2 weeks of blinded treatment to taper off study drug treatment. The assignment will be done by a computer generated system and neither the trial doctor or the participant or their caregivers will know which treatment is being given to them. The dose of the treatment will depend on the weight of the participants. If the participants weigh less than or equal to 35 kg, they will receive 2 sachets of the gel twice a day (1 sachet approximately every 12 hours) and if they weigh more than 35 kg, they will receive 4 sachets of gel per day (2 sachets approximately every 12 hours). Parents/ caregivers will be instructed on proper application of the gel. The gel will be applied to clean, dry, intact skin of the upper arms/ shoulders.

Blood samples will be collected for safety analysis of ZYN002. An independent analytical laboratory will also perform CGG repeat and methylation status analyses. Additionally, the parents/caregivers will be asked to complete some questionnaires. There will be other questionnaires and scales that will be completed at the site by the trial doctor.

After the final dose, patients will be followed weekly for 4 weeks by telephone, prior to discharge from the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children and adolescents aged 3 to less than 18 years, at the time of Screening.
* Diagnosis of FXS through molecular documentation of FMR1 full mutation.
* Judged to be in good health based on physical exam, 12-lead ECG and clinical laboratory test results.
* Patients must be assessed by the Investigator as being moderately to severely impacted due to FXS.
* Patients taking psychotropic medication(s) should be on a stable regimen of not more than two such medications for at least fours weeks preceding Screening and must maintain that regimen throughout the study.
* If patients are receiving non-pharmacological, behavioral and/or dietary interventions, they must be stable and have been doing so for three months prior to screening.
* Patients and parents/caregivers must be adequately informed of the nature and risks of the study and given written informed consent prior to Screening.
* In the Investigator's opinion, patients and parents/caregivers are reliable and willing and able to comply with all protocol requirements and procedures.

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy.
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or total bilirubin levels greater than or equal to 2 times the upper limit of normal or alkaline phosphatase levels greater than or equal to 3 times the upper limit of normal.
* Use of a strong inhibitor/inducer of CYP3A4 or sensitive substrate of CYP3A4.
* Use of minocycline for 30 days prior to screening or throughout the study.
* Use of any benzodiazepine at screening or throughout the study.
* Use of THC or CBD-containing product within three months of Screening Visit or during the study.
* Change in pharmacologic or non-pharmacologic intervention during the course of the study.
* Any skin disease or condition including eczema, psoriasis, melanoma, acne, contact dermatitis, scarring, imperfections, lesions, tattoos, or discoloration that may affect treatment application, application site assessments or absorption of the trial drug.
* Patient is using the following ASMs: clobazam, phenobarbital, ethosuximide, felbamate or vigabatrin.
* Patients has an advanced, severe or unstable disease that may interfere with the study outcome evaluations.
* Patient has acute or progressive neurological disease, psychosis, schizophrenia or any other psychiatric disorder or severe mental abnormalities (other than FXS) that are likely to require changes in drug therapy or interfere with the study objectives or ability to adhere to protocol requirements.
* Patient has suspected or confirmed cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, cardiac conduction problems, exercise-related cardiac events including syncope and pre-syncope, risk factors for Torsades de pointes (e.g. heart failure, hypokalemia, family history of Long QT Syndrome) or other serious cardiac problems.
* History of treatment for, or evidence of drug abuse within the past year.
* Patient responds "yes" to Question 4 or 5 on the C-SSRS (Children) during Screening or at any time on study.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (17):
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - UC Davis Health System, MIND Institute, Sacramento, California
  - Children's Hospital of Colorado, Denver, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Fragile X Center of Atlantic Health System, Morristown, New Jersey
  - The Fragile X Spectrum Disorder Clinic at Icahn School of Medicine at Mount Sinai, Division of Medical Genetics, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Central States Research, Tulsa, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Greenwood Genetic Center, Greenville, South Carolina
  - University of Washington Center for Human Development and Disability, Seattle, Washington
- Australia (3):
  - Westmead Children's Hospital, Sydney, New South Wales
  - Lady Cilento Children's Hospital - South Brisbane, Brisbane, Queensland
  - Genetics Clinics Australia, Melbourne, Victoria
- Wellington Hospital, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berry-Kravis E, Hagerman R, Budimirovic D, Erickson C, Heussler H, Tartaglia N, Cohen J, Tassone F, Dobbins T, Merikle E, Sebree T, Tich N, Palumbo JM, O'Quinn S. A randomized, controlled trial of ZYN002 cannabidiol transdermal gel in children and adolescents with fragile X syndrome (CONNECT-FX). J Neurodev Disord. 2022 Nov 25;14(1):56. doi: 10.1186/s11689-022-09466-6. PMID 36434514
- [Derived] Heussler HS. Emerging Therapies and challenges for individuals with Angelman syndrome. Curr Opin Psychiatry. 2021 Mar 1;34(2):123-128. doi: 10.1097/YCO.0000000000000674. PMID 33395098

RESULTS

PARTICIPANT FLOW:
Groups:
- ZYN002 - Cannabidiol Transdermal Gel: ZYN002 supplied as a transdermal gel. Patients weighing less than or equal to 35 kg will be randomized to receive either 125 mg cannabidiol Q12H or placebo.
  Patients weighing greater than 35 kg will be randomized to receive 250 mg cannabidiol Q12H or placebo.
  ZYN002 - Cannabidiol Transdermal Gel: Pharmaceutically manufactured. Cannabidiol formulated as a clear gel (transdermal delivery)
Period: Overall Study
Arm/Group | ZYN002 - Cannabidiol Transdermal Gel | Placebo Transdermal Gel
Started | 110 | 102
Completed | 106 | 99
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZYN002 - Cannabidiol Transdermal Gel | Placebo Transdermal Gel | Total
Number analyzed (Participants) | 110 | 102 | 212
Age, Continuous [Mean (Full Range); unit: years] | 9.6 [3 to 17] | 9.8 [3 to 17] | 9.7 [3 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 53
  Male | 81 | 78 | 159
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 7 | 4 | 11
  White | 85 | 81 | 166
  More than one race | 6 | 7 | 13
  Unknown or Not Reported | 9 | 5 | 14
ABC-C FXS [Mean (Standard Deviation); unit: units on a scale] — Population: One participant did not receive trial medication and one patient did not have a post-baseline efficacy measure, resulting in 210 participants in the full analysis set (ZYN002: n=109); placebo: n=101).
  units on a scale
    Social Avoidance Subscale: number analyzed (Participants) | 109 | 101 | 210
    Social Avoidance Subscale | 7.12 (2.71) | 7.24 (2.80) | 7.18 (2.75)
    Irritability Subscale: number analyzed (Participants) | 109 | 101 | 210
    Irritability Subscale | 28.49 (13.10) | 27.65 (12.96) | 28.09 (13.01)
    Socially Unresponsive / Lethargic: number analyzed (Participants) | 109 | 101 | 210
    Socially Unresponsive / Lethargic | 13.42 (6.75) | 12.82 (7.09) | 13.13 (6.90)

OUTCOME MEASURES:

1. Primary Outcome: Aberrant Behavior Checklist-Community Fragile X Factor Structure (ABC-C FXS) Social Avoidance Subscale - Full Analysis Set
Description: The Aberrant Behavior Checklist-Community is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials. The range for score for the subscale is from 0 to 12, and a higher value indicates a worse outcome.
Time Frame: Change from Baseline to end of treatment (Week 12)
Population: The prospective comparison of the full analytical set between ZYN002 and placebo.
Measure: Least Squares Mean (Standard Error); unit: change in score
Groups:
- Placebo: Placebo formulated as a clear gel (transdermal delivery)
Arm/Group | ZYN002 - Cannabidiol Transdermal Gel | Placebo
Number analyzed (Participants) | 109 | 101
change in score | -2.68 (0.310) | -2.29 (0.318)
Statistical Analysis 1: Comparison: ZYN002 - Cannabidiol Transdermal Gel vs Placebo; Test type: Superiority; p = 0.321, MMRM - Mixed model for repeated measures

2. Secondary Outcome: Aberrant Behavior Checklist-Community Fragile X Factor Structure (ABC-C FXS) Irritability Subscale - Full Analysis Set
Description: The Aberrant Behavior Checklist-Community is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials. The range for score for the subscale is between 0 and 54, and the higher score means a worse outcome.
Time Frame: Change from baseline to end of treatment (Week 12)
Population: The prospective comparison of the full analytical set between ZYN002 and placebo.
Measure: Least Squares Mean (Standard Error); unit: Change in score
Arm/Group | ZYN002 - Cannabidiol Transdermal Gel | Placebo Transdermal Gel
Number analyzed (Participants) | 109 | 101
Change in score | -5.88 (0.960) | -4.14 (0.984)
Statistical Analysis 1: Comparison: ZYN002 - Cannabidiol Transdermal Gel vs Placebo Transdermal Gel; Test type: Superiority; p = 0.149, MMRM - Mixed model for repeated measures

3. Secondary Outcome: Aberrant Behavior Checklist-Community, Fragile X Factor Structure (ABC-C FXS) Socially Unresponsive/Lethargic Subscale - Full Analysis Set
Description: The Aberrant Behavior Checklist-Community is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials. The range for score for the subscale is from 0 and 39, and a higher mean indicates a worse outcome.
Time Frame: Change from baseline to end of treatment (Week 12)
Population: The prospective comparison of the full analytical set between ZYN002 and placebo.
Measure: Least Squares Mean (Standard Error); unit: Change in score
Arm/Group | ZYN002 - Cannabidiol Transdermal Gel | Placebo Transdermal Gel
Number analyzed (Participants) | 109 | 101
Change in score | -3.50 (0.565) | -3.14 (0.577)
Statistical Analysis 1: Comparison: ZYN002 - Cannabidiol Transdermal Gel vs Placebo Transdermal Gel; Test type: Superiority; p = 0.607, MMRM - Mixed model for repeated measures

4. Secondary Outcome: Number of Participants With Any Improvement - Clinical Global Impressions- Improvement (CGI-I) - Full Analysis Set
Description: The Clinical Global Impressions- Improvement global improvement item is a 7-point Likert scale designed to measure behavioral symptomatic change at a specific time compared to baseline. CGI-I is a standard global measure of potential change with treatment in placebo-controlled pharmacotherapy trials in developmental disabilities. The score ranges form 1-very much improved to 7-very much worse. The percentage of patients with any improvement (minimally, much, very much improved) was assessed.
Time Frame: Change in CGI-I at end of treatment (Week 12)
Population: The prospective comparison of the full analytical set between ZYN002 and placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | ZYN002 - Cannabidiol Transdermal Gel | Placebo Transdermal Gel
Number analyzed (Participants) | 109 | 101
Participants | 46 | 37
Statistical Analysis 1: Comparison: ZYN002 - Cannabidiol Transdermal Gel vs Placebo Transdermal Gel; Test type: Superiority; p = 0.426, ANOVA

5. Primary Outcome: Aberrant Behavior Checklist-Community Fragile X Factor Structure (ABC-C FXS) Social Avoidance Subscale - Ad Hoc Analysis
Description: The Aberrant Behavior Checklist-Community is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials. The range for score for the subscale is from 0 and 12, and the higher score means a worse outcome.
Time Frame: Change from baseline to end of treatment (Week 12)
Population: A pre-specified, ad hoc analysis of the data collected in patients with ≥90% methylation of the FMR1 gene to evaluate the effect of ZYN002 versus placebo was developed prior to unblinding the trial.
Measure: Least Squares Mean (Standard Error); unit: Change in score
Arm/Group | ZYN002 - Cannabidiol Transdermal Gel | Placebo
Number analyzed (Participants) | 91 | 76
Change in score | -2.99 (0.323) | -1.99 (0.345)
Statistical Analysis 1: Comparison: ZYN002 - Cannabidiol Transdermal Gel vs Placebo; Test type: Superiority; p = 0.02, MMRM - Mixed model for repeated measures

6. Secondary Outcome: Aberrant Behavior Checklist-Community Fragile X Factor Structure (ABC-C FXS) Irritability Subscale - Ad Hoc Analysis
Description: as for outcome 2
Time Frame: Change from baseline in ABC-C to end of treatment (Week 12)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Change in score
Arm/Group | ZYN002 - Cannabidiol Transdermal Gel | Placebo Transdermal Gel
Number analyzed (Participants) | 91 | 76
Change in score | -6.43 (1.020) | -4.13 (1.088)
Statistical Analysis 1: Comparison: ZYN002 - Cannabidiol Transdermal Gel vs Placebo Transdermal Gel; Test type: Superiority; p = 0.091, MMRM - Mixed model for repeated measures

7. Secondary Outcome: Aberrant Behavior Checklist-Community Fragile X Factor Structure (ABC-C FXS) Socially Unresponsive/Lethargic Subscale - Ad Hoc Analysis
Description: The Aberrant Behavior Checklist-Community is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials. The range for score for the subscale is from 0 to 39 , and the higher score means a worse outcome.
Time Frame: Change from baseline in ABC-C to end of treatment (Week 12)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Change in score
Arm/Group | ZYN002 - Cannabidiol Transdermal Gel | Placebo Transdermal Gel
Number analyzed (Participants) | 91 | 76
Change in score | -3.91 (0.592) | -2.74 (0.631)
Statistical Analysis 1: Comparison: ZYN002 - Cannabidiol Transdermal Gel vs Placebo Transdermal Gel; Test type: Superiority; p = 0.135, MMRM - Mixed model for repeated measures

8. Secondary Outcome: Number of Participants With Any Improvement - Clinical Global Impressions- Improvement (CGI-I) - Ad Hoc Analysis
Description: as for outcome 4
Time Frame: Change in CGI-I at end of treatment (Week 12)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ZYN002 - Cannabidiol Transdermal Gel | Placebo Transdermal Gel
Number analyzed (Participants) | 91 | 76
Participants | 43 | 25
Statistical Analysis 1: Comparison: ZYN002 - Cannabidiol Transdermal Gel vs Placebo Transdermal Gel; Test type: Superiority; p = 0.056, MMRM - Mixed model for repeated measures

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 18 weeks.
Description: Adverse Event Analysis Population Description: 212 patients (ZYN002: n=110; placebo: n=102) were enrolled in the study. One participant did not receive trial medication and is excluded from the safety population, resulting in 211 participants included in safety analysis (ZYN002: n=109); placebo: n=102).
Arm/Group | ZYN002 - Cannabidiol Transdermal Gel | Placebo Transdermal Gel
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/102
Other Adverse Events (participants affected / at risk) | 45/109 | 30/102
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZYN002 - Cannabidiol Transdermal Gel (N=109) | Placebo Transdermal Gel (N=102)
vomiting (Gastrointestinal disorders) | 8 (9) | 6 (7)
pyrexia (General disorders) | 5 (5) | 7 (7)
application site pain (General disorders) | 7 (7) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 15 (16) | 7 (7)
nasopharyngitis (Infections and infestations) | 10 (10) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT03614663/Prot_SAP_000.pdf